CLINICAL TRIAL: NCT04655859
Title: Evaluation of Saliva Thiol/Disulfide Homeostasis and Oxidative Stress in Children With Severe Early Childhood Caries by a Novel Method- Part 1
Brief Title: Thiol/Disulfide and Oxidative Stress
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aslı Sogukpınar, Dr., Kahramanmaras Sutcu Imam University
Other Study IDs: 2020/1-19M
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Severe Early Childhood Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- severe early childhood caries
  Interventions: Diagnostic Test: saliva cotton swab
- healthy children
  Interventions: Diagnostic Test: saliva cotton swab

INTERVENTIONS:
Diagnostic Test: saliva cotton swab — evaluate the role of thiol/disulfide homeostasis and oxidative stress in the saliva of children with severe early childhood caries and healthy group

SUMMARY:
The aim of this study was to evaluate the role of thiol/disulfide homeostasis and oxidative stress in the saliva of children with severe early childhood caries

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years

Exclusion Criteria:

* the children with systemic illness, using anti-inflammatory drug

Ages: 3 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: the children with severe early childhood caries which are 3-5 years
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
thiol/disulfide homeostasis | six months
  Unstimulated saliva samples were taken from all children. Then, thiol/disulfide homeostasis and antioxidant levels were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Soğukpınar, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The thiol/disulfide homeostasis and antioxidant levels is to be shared in this study.